CLINICAL TRIAL: NCT00904631
Title: A Prospective, Open Label, Non Randomized, Clinical Study to Evaluate the Safety and Effectiveness of the Eraser Tattoo Removal Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Ori Nesher, Hawk Medical Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 33/08
Record Dates: First submitted 2009-05-19; First posted 2009-05-20 (Estimated); Last update posted 2009-05-20 (Estimated); Status verified 2009-05

CONDITIONS: Removal of Colors Tattoo (Multiple Colors)

ARMS (1):
- Treatment (Experimental): Subjects will be treated with the Eraser device, using salicylic acid (5%) as washing fluid. The skin will be examined by a physician and the tattoo area will be photographed. The Eraser device will be used to remove the tattoo from the entire tattoo area (up to 30 minutes in a single session). An absorbent bandage will be put on the treated area for one-hour post treatment. After Care Treatment, based on a Dermatologist's consultation, will be performed on a case-by-case basis (for example, use of antibiotic ointments in case of infection).
  Interventions: Device: Eraser device+ salicylic acid (5%)

INTERVENTIONS:
Device: Eraser device+ salicylic acid (5%) — Subjects will be treated with the Eraser device, using salicylic acid (5%) as washing fluid. The skin will be examined by a physician and the tattoo area will be photographed. The Eraser device will be used to remove the tattoo from the entire tattoo area (up to 30 minutes in a single session). An absorbent bandage will be put on the treated area for one-hour post treatment. After Care Treatment, based on a Dermatologist's consultation, will be performed on a case-by-case basis (for example, use of antibiotic ointments in case of infection).

SUMMARY:
Name of Device: Eraser Tattoo Removal Device

Device Description: The Eraser device is a mechanical device, resembling tattoo devices but with an innovative mechanism for dripping treatment fluid over reciprocating needles and returning used fluid into a reservoir chamber. The device is intended for removal of tattoos.

Objectives: This study is a continuation of a previous feasibility study, which tested the ability of the device to remove tattoos from small skin areas. The purpose of this study is to evaluate the safety and effectiveness of the Eraser Tattoo Removal system for removal of skin tattoos in their entirety.

Subject Population: 20 patients in the medical center. Subject enrollment will include (i) a variety of tattoo colors (multiple colors) (ii) a variety of tattoo composition, contour lines and shadings (iii) Subjects with different skin colors (white, tanned, dark, etc…) (iv) professional and amateur tattoos.

Structure: A prospective, non-randomized, open, clinical study designed according to FDA guidelines; ISO 14155: standard for clinical studies of medical devices; and the procedures of the Israeli Ministry of Health for clinical studies.

After informed consent is signed, demographic details and medical history will be taken and a physical examination performed. Subjects will be treated with the Eraser device, using salicylic acid (5%) as washing fluid. The skin will be examined by a physician and the tattoo area will be photographed. The Eraser device will be used to remove the tattoo from the entire tattoo area (up to 30 minutes in a single session). An absorbent bandage will be put on the treated area for one-hour post treatment. After Care Treatment, based on a Dermatologist's consultation, will be performed on a case-by-case basis (for example, use of antibiotic ointments in case of infection). All subjects must refrain from exposure to the sun for 90 days following each treatment.

Follow-up: The subject will return for follow-up at one week, two weeks, 1 month and two months (if tattoo removal and skin healing is complete), or up to six months (if skin healing/ tattoo removal are not complete by two months), or until the healing of the tattoo removal site is completely resolved or until the investigator determines that additional treatments will provide no further benefit to the patient. In each follow-up visit, a physician will perform a physical examination, check the skin over and around the treatment area, and take photographs of the treated area. Images from last follow-up will be compared with images of the same site taken before the removal procedure, for evaluation of treatment efficacy and safety.

Repeat treatments: if tattoo removal is not complete, up to two additional treatments will be performed, based on the investigator's discretion. After each treatment, follow-up will continue as described above.

Blinding: Non-Applicable Concurrent Control: There is no concurrent control group in this study. Images of tattoos before treatment will serve as the reference measure, to which images of healed skin, several weeks after tattoo removal, will be compared.

Sample Size: 20 subjects will be enrolled in the study. Primary Effectiveness Variables: The primary measure of effectiveness will be the pigment clearance, as evaluated by image comparison on a 1-5 analog scale (5 - 81-100% clearance- excellent removal; 4 - 61-80% - good removal; 3 - 41-60% - moderate removal; 2 - 21-40% - fair removal; 1 - 0-20% - poor removal). Effectiveness will be calculated for the total study group and for individual sub-groups (skin type, pigment colors, etc.). Effectiveness will be analyzed separately for the area affected (percentage of treated area that showed any reaction to treatment) and for the change in color brightness (if, due to technical reasons, part of the tattoo showed a major effect, this area will be evaluated for the change in color brightness). For both analyses, the same scale will be used.

For safety assessment, the rate of systemic and dermatologic adverse events will be calculated and reported. The data will be listed by type of event and by severity. Specifically, textural change, hypo- and hyper- pigmentation will be followed and their rates calculated.

Data Analysis: For this clinical study, descriptive statistics will be used. Successful treatment will be a result of 3 or more (at least, moderate tattoo removal) on the brightness change scale.

Study Sponsor: Hawk Medical Technologies Ltd.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 years or older, of any race.
2. Subject has a tattoo for removal on the back, shoulders or abdomen (areas that can usually be hidden).
3. Subjects willing to participate as evidenced by signing the written informed consent.

Exclusion Criteria:

1. Subject has a dermatological disease, active or latent (e.g. psoriasis)
2. Subject has a known tendency for Keloid formation.
3. Subject has a known tendency for skin hyperpigmentation.
4. Subject is susceptible to Koebner reaction.
5. Subject has blood transmittable diseases (HIV, HBV, HCV, etc.)
6. Subject has known allergy to device components/ treatment fluids (stainless steel for needles; salicylic acid; aspirin; K-Y gel).
7. Subject has medical conditions that may be worsened by concomitant use of aspirin (Hematologic, renal, GI, hepatic or gastrointestinal contraindications; viral illness or fever; old age increases susceptibility to toxic effects); topical salicylic acid (condylomata acumynata, open wounds, burns, diabetes mellitus, peripheral vascular disease, skin and skin structure infections, skin inflammation, skin irritation) or worsened by local anesthesia materials.
8. Subject is taking aspirin or anti-coagulant medications; or using topical salicylic acid preparations.
9. Female subject who is pregnant or lactating.
10. Subject participates in any other clinical study at the same time

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-05 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
For this clinical study, descriptive statistics will be used. Successful treatment will be a result of 3 or more (at least, moderate tattoo removal) on the brightness change scale. | two months

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf-Harofeh Medical Center, Ẕerifin, Israel